CLINICAL TRIAL: NCT03320031
Title: A Randomized, Open, Controlled, Parallel Group Study of Adding Linagliptin to Control Glycemic Variability and HbA1c in Peritoneal Dialysis Patients With Type 2 Diabetes(PDPD) With Premixed Insulin Therapy
Brief Title: A Study of Adding Linagliptin to Control Glycemic Variability and HbA1c in Peritoneal Dialysis Patients With Type 2 Diabetes(PDPD) With Premixed Insulin Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanbing Li (Other)
Responsible Party: Sponsor-Investigator, Yanbing Li, Director of Endocrinology and Metabolism Department, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017187
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus; Peritoneal Dialysis
Keywords: Linagliptin; premixedinsulin therapy; peritoneal dialysis; glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; insulin lispro, isophane insulin lispro drug combination (25:75)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined group (Experimental): Drug: linagliptin&premixed insulin Treated with linagliptin 5mg/d combined with premixed insulin for 12 weeks.
  Interventions: Drug: Linagliptin; Drug: Humalog Mix 75/25
- linsulin group (Active Comparator): Drug: premixed insulin Treated with premixed insulin for 12 weeks.
  Interventions: Drug: Humalog Mix 75/25

INTERVENTIONS:
Drug: Linagliptin — Take linagliptin 5mg a day.
  Other Names: Trajenta
  Arms: combined group
Drug: Humalog Mix 75/25 — Administer subcutaneous premixed insulin twice a day.
  Other Names: insulin lispro 75/25

SUMMARY:
In china, there are the most population of type 2 diabetes mellitus (DM) among the world and DM becomes currently the second cause for end-stage renal disease (ESRD). Nearly 50% of insulin-treated PD patients in clinical practice are treated with premixed insulin. Glycemic control in them is very difficult to be achieved mainly due to the uremic status of these patients and glucose exposure from peritoneal dialysate, a higher glycemic variability and higher risk of hypoglycemia. Linagliptin, unlike other DPP-4 inhibitors, has a primarily non-renal elimination route, and does not require dose adjustment for any level of impaired renal function. The aim of this study is to evaluate the effect of linagliptin on glucose variability and glycemic control in peritoneal dialysis patients with type 2 diabetes who are inadequately controlled with premixed insulin therapy.

This will be a randomized, double-blind, placebo-controlled, parallel group study to evaluate the effect of linagliptin on glucose variability and glycemic control in peritoneal dialysis patients with type 2 diabetes who are inadequately controlled with premixed insulin therapy.which will be conducted in 8 diabetes centres and/or nephropathy departments in China. After a 4-week run- in period, 232 participants are randomized (1:1) to either premixed insulin combined with linagliptin (5mg/d) group (also named combined group) or premixed insulin alone group (also named insulin group) for 12 weeks. Finally, the primary endpoint is glucose variability indicated by MAGE, secondary endpoints include HbA1c, FPG, PPG, LAGE, SDBG, PT10.0, PT3.9, 1h fasting MBG, 3h postprandial MBG, insulin dosage, hypoglycemia and body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients who were treated with insulin regimen;
2. Ages eligible for study:18 years to 80 years;
3. The patients with end-stage kidney disease receiving a regular peritoneal dialysis for at least 3 months;
4. HbA1c ranging from 6.5%-10.5% when screening and randomizing ;
5. Body mass index ranging from 21 to 35 kg/m2.

Exclusion Criteria:

1. Having any severe acute or chronic diabetic complications
2. Blood aminotransferase level rising up more than 2 times of the upper normal limit
3. Any severe cardiac disease, severe systemic diseases or malignant tumour
4. Female patients incline to be pregnant
5. Being treated with corticosteroid, immunosuppressing drugs or cytotoxic drugs
6. Poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2017-06-03 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
glucose variability | 12 weeks
  The change from baseline to week 12 in glucose variability indicated by MAGE.

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  Changes in HbA1c between two groups
FPG | 12 weeks
  Changes in FPG between two groups
insulin dosage | 12 weeks
  Changes in FPG at the end between two groups
body weight | 12 weeks
  Changes in body weight at the end between two groups
hypoglycemia | 12 weeks
  Frequency of hypoglycemia at the end in each gropu

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China